CLINICAL TRIAL: NCT05447988
Title: Post-Marketing Clinical Follow-Up Study to Confirm the Safety and Effectiveness/Performance of Motiva Flora® Tissue Expander in Staged Breast Reconstruction Surgery
Brief Title: Motiva Flora Tissue Expander PMCF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Establishment Labs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLINP-001001
Record Dates: First submitted 2021-07-23; First posted 2022-07-07 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Breast Tissue Accessory; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Tissue Expansion Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Two-stage reconstruction (Other): 136 participants will undergo two-stage reconstruction
  Interventions: Device: Breast Tissue Expander

INTERVENTIONS:
Device: Breast Tissue Expander — tissue expander based breast reconstruction
  Other Names: Motiva Flora Tissue Expander

SUMMARY:
The Motiva Flora® Tissue Expander clinical study (hereafter Motiva Flora® TE study) is a 6-month, open-label, prospective, multicentre post-marketing follow-up study designed to confirm the Safety and Effectiveness/Performance of Motiva Flora® TE in breast reconstruction surgery.

The study will include 136 women, planned for staged breast reconstruction, in 6 countries (Spain, Belgium, France, Costa Rica, Chile and Panama). Breast tissue expansion and the final breast implant will be performed using devices from the Motiva Flora® TE catalogue.

ELIGIBILITY:
Inclusion Criteria

* The participant gives written informed consent.
* The participant is genetically female, aged 18 years or older.
* The participant needs tissue expansion as part of breast reconstruction treatment following mastectomy, which may include immediate reconstruction.
* The participant is in a suitable clinical condition to allow breast implant placement after tissue expander placement, at the discretion of the investigator.
* The participant has the physical and cognitive capacity to understand and follow the surgeon's recommendations.
* Complete radiotherapy at least 1 year before surgery.
* Partial or total decrease in tumour volume after radiotherapy.
* The participant is able and willing to comply with all study requirements including attending follow-up appointments.
* Participant with reasonable surgical risk.
* Participant with a history of non-metastatic breast cancer.
* Participant willing to undergo an MRI, CT scan and any other studies if required at surgeon discretion.

For substudy - MRI / CT - the following additional criteria apply:

- Patient is willing to undergo one MRI and one CT anytime during the follow up

Exclusion Criteria:

* The participant is pregnant or planning a pregnancy during the first year after surgery or is currently breastfeeding.
* Participants with implanted devices that may be affected by magnetic fields (pacemakers, drug infusion devices).
* Participants with abnormal haematological and biochemical values after chemotherapy.
* Participants with tumour residues in or near the area where tissue expansion is to be performed.
* Participants who do not have adequate tissue at the intended site for expansion, at the surgeon's discretion, due to previous radiotherapy, ulceration, vascular involvement, history of impaired wound healing or scar deformity.
* Participants with current or previous infection in the area where the expansion will take place.
* Presence of autoimmune diseases such as lupus or scleroderma, or immunocompromised participants due to immunosuppressive or steroid therapy.
* Inadequate chest wall tissue due to damage caused by radiotherapy, tight skin grafts or radical resection of the pectoralis major muscle.
* Participant who is included in another pharmacological or device research study.
* Participants with a previous history of failure of attempted tissue expansion or breast implant placement at the site of intended expansion.
* Participant with a history of silicone sensitivity.
* Employees of Establishment Labs or any of its divisions or sites; Researchers or anyone who collaborates on the study or is directly related to a person working for Establishment Labs, sites or commissioned Researchers.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2020-12-14 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of the device and procedure-related adverse events | 6 months follow-up
  Cumulative incidence of the device and procedure-related adverse events as assessed by occurrence, seriousness, severity, causal relationship with the device
Perceived success of breast tissue expansion | 6 months follow-up
  Success of the process as perceived by the investigator considering change in final breast volume and comparison with expected volume
Expected completion of breast tissue expansion | Up to 6 months follow-up
  Evaluate the time it took to reach the desired expansion following planning.
Satisfaction assessed by the 5 point Likert scale | 6 months follow-up
  - Surgeon's overall satisfaction (1=very significant improvement, 2=significant improvement, 3=improvement, 4=no change and 5=decline) at each follow-up visit.

SECONDARY OUTCOMES:
Integrity of the fixing tabs defined as tabs being intact at explantation | During the intervention/procedure/surgery for explantation
  Observation of Integrity of the fixing tabs defined as tabs being intact at explanation with no detachments and cuts.
MRI and potential incidents | Up to 6 months follow-up
  Incidents attributable to MR exposure.
MRI and port locator performance measured through accurate locator function | Up to 6 months follow-up
  Motiva Flora® Port locator performance after MRI measured through accurate location defined when the green light on the device comes on
Device interference on MRI | Up to 6 months follow-up
  Device interference on MRI measured through artifact size
In vivo testing of device interference with CT radiotherapy planning. | Up to 6 months follow-up
  Radiological Report after undergo CT:
  - Interference with CT.

CONTACTS AND LOCATIONS:
Locations (5):
- Centro de Cirugía Plástica y Reconstructiva. Dra. Viviana Spröhnle Hospital Regional de Rancagua, Rancagua, Chile
- Centro Europeo de Cirugia, San José, Provincia de San José, Costa Rica
- The Panama Clinic Complejo Hospitalario Pacific Center, Panama City, Panama
- Spain (2):
  - Centro de Patología de la Mama, Madrid
  - Hospital Gregorio Marañón, Madrid

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://motiva.health